CLINICAL TRIAL: NCT07366073
Title: A Randomized Two-Group Pretest-Posttest Study of Virtual Reality-Based Dementia Education Among College Students
Brief Title: Effects of Virtual Reality Dementia Education on College Students' Knowledge and Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC113-09
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Dementia Education
Keywords: Virtual reality; Dementia education; College students; Attitudes toward dementia; Health education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of two parallel groups and received a single type of virtual reality-based dementia education (VR-360 or computer-generated VR) throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR-360 Group (Experimental): Participants in this arm received a virtual reality 360-degree (VR-360) dementia education intervention based on immersive real-life video scenarios designed to improve dementia-related knowledge and attitudes.
  Interventions: Other: VR-360 Dementia Education
- CG-VR Group (Experimental): Participants in this arm received a computer-generated virtual reality (CG-VR) dementia education intervention delivered through an interactive virtual learning environment to enhance dementia-related knowledge and attitudes.
  Interventions: Other: CG VR Dementia Education

INTERVENTIONS:
Other: VR-360 Dementia Education — An immersive virtual reality 360-degree educational program designed to improve dementia-related knowledge and attitudes through real-life video scenarios.
  Arms: VR-360 Group
Other: CG VR Dementia Education — A computer-generated virtual reality educational program designed to enhance dementia-related knowledge and attitudes using an interactive virtual learning environment.
  Arms: CG-VR Group

SUMMARY:
Dementia is a growing public health concern, and improving knowledge and attitudes toward dementia is important for reducing stigma and promoting supportive care. Virtual reality (VR) has been increasingly used as an educational tool because it can provide immersive and engaging learning experiences.

The purpose of this study is to examine the effects of different types of virtual reality-based dementia education on college students' knowledge of dementia and their attitudes toward people living with dementia. College students were randomly assigned to one of two educational approaches: a VR-360 experience based on real-life scenarios or a computer-generated VR (CG-VR) learning environment.

Participants completed questionnaires assessing dementia-related knowledge and attitudes before and after the educational intervention. By comparing changes between the two groups, this study aims to determine whether different VR formats lead to different learning outcomes. The findings of this study may help inform the design of future dementia education programs using immersive technologies.

DETAILED DESCRIPTION:
This study adopted a two-group randomized pretest-posttest design to evaluate the effectiveness of different virtual reality-based dementia education approaches. Participants were recruited from a university in central Taiwan and were randomly assigned to either a VR-360 group or a computer-generated VR (CG-VR) group using computer-generated random codes.

Both interventions were designed to introduce key concepts related to dementia, including common warning signs, prevention strategies, and communication considerations when interacting with people living with dementia. The VR-360 intervention used immersive real-life video scenarios, whereas the CG-VR intervention used a virtual learning environment with interactive instructional content.

Dementia-related knowledge and attitudes were assessed using standardized questionnaires before and after the intervention. Changes in outcomes were compared between groups to evaluate the differential effects of the two VR formats. This study was approved by the Institutional Review Board of Taichung Tzu Chi Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 20 years and older.
* College students who are able to participate in virtual reality-based teaching activities and complete questionnaire assessments.
* Willingness to participate and provide written informed consent.

Exclusion Criteria:

* Individuals with visual or auditory impairments that may interfere with virtual reality use.
* Individuals with abnormalities of the head or face that prevent wearing virtual reality equipment.
* Individuals who are unable to adapt to virtual reality devices (e.g., experiencing severe motion sickness).

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Attitudes Toward Dementia | Baseline (pre-intervention) and immediately after the intervention
  Attitudes toward dementia were measured using a self-administered questionnaire before and after the intervention.
Dementia Knowledge | Baseline (pre-intervention) and immediately after the intervention
  Dementia-related knowledge was assessed using a structured questionnaire before and after the virtual reality-based educational intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University in Central Taiwan, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No